CLINICAL TRIAL: NCT02272374
Title: Vascular Access Choice and Outcomes in the Elderly and Very Elderly With End Stage Renal Disease in China :a Multicenter Prospective Cohort Study
Brief Title: Vascular Access Choice and Outcomes in the Elderly and Very Elderly With End Stage Renal Disease in China
Acronym: ACCESS-China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director, Division of Nephrology, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZHKI-HDVA-004
Record Dates: First submitted 2014-09-23; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Arteriovenous fistula; Tunneled cuffed catheter; Arteriovenous graft; Elderly; Very elderly
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- e-AVF group (Experimental): 120 elderly with end stage renal disease will undergo AVF creation.
  Interventions: Procedure: AVF creation
- e-TCC group (Experimental): 120 elderly with end stage renal disease will undergo TCC placement.
  Interventions: Procedure: TCC placement
- e-AVG group (Experimental): 60 elderly with end stage renal disease will undergo AVG creation.
  Interventions: Procedure: AVG creation
- ve-AVF group (Experimental): 80 very elderly with end stage renal disease will undergo AVF creation.
  Interventions: Procedure: AVF creation
- ve-TCC group (Experimental): 80 very elderly with end stage renal disease will undergo TCC placement.
  Interventions: Procedure: TCC placement
- ve-AVG group (Experimental): 40 very elderly with end stage renal disease will undergo AVG creation.
  Interventions: Procedure: AVG creation

INTERVENTIONS:
Procedure: AVF creation
  Other Names: Arteriovenous fistula creation
  Arms: e-AVF group; ve-AVF group
Procedure: TCC placement
  Other Names: Tunneled cuffed catheter placement
  Arms: e-TCC group; ve-TCC group
Procedure: AVG creation
  Other Names: Arteriovenous graft creation
  Arms: e-AVG group; ve-AVG group

SUMMARY:
The purpose of the study is to evaluate the clinical outcomes and cost-effectiveness of different vascular access(arteriovenous fistula, tunneled cuffed catheter and arteriovenous graft) in the elderly and very elderly with end-stage renal disease in China.

ELIGIBILITY:
Inclusion Criteria:

1. The elderly and very elderly with end stage renal disease.
2. Estimated glomerular filtration rate (eGFR) <20ml/min*1.73m2
3. All study subjects agree to participate in the study and provide written informed consent.

Exclusion Criteria:

1. Patients' life expectancy is less than 2 years.
2. Mental illness that makes the patients unable to complete the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The patency rate of vascular access | 2 years
  Including primary and secondary patency rate.Blood flow can be above 500 mL/min in a mature arteriovenous fistula by ultrasound scan and 4 times of body weight (Kg*4 mL/min) in a arteriovenous graft or tunneled cuffed catheter in dialysis practice.
Effect of vascular access construction on ventricular volumes and left ventricular remodeling | 2 years
  Assessed by doppler echocardiography
Effect of vascular access construction on brain MRI and cognitive functionslesions and cognitive function | 2 years
  Cognitive functions are assessed by psychic and autonomy scores

SECONDARY OUTCOMES:
Complications of vascular access | 2 years
  Described as %.Complications including bleeding, infection, thrombosis, artery steal syndrome, heart failure, inadequate dialysis, etc.
Cost-effectiveness of different vascular access | 2 years
  Described as $.The cost including medical expenses and non-medical expenses.
Hospitalization rate due to vascular access. | 2 years
Mortality due to vascular access | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, master, Principal Investigator — Division of Nephrology, Shanghai ChangZheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China